CLINICAL TRIAL: NCT02028936
Title: Study of the Impact of the Regular Consumption of Polyphenol-rich Grape Juice on the Biological Parameters of Oxidative Stress and on Endothelial Function in Healthy Subjects: a Prospective Randomised Double-blind Study
Brief Title: Study of the Impact of the Regular Consumption of Polyphenol-rich Grape Juice on the Biological Parameters of Oxidative Stress and on Endothelial Function in Healthy Subjects
Acronym: Fijus Raisol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: BARDOU FUI 2013
Record Dates: First submitted 2013-12-18; First posted 2014-01-07 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Healthy Subjects

ARMS (2):
- Grape juice rich in polyphenols (Experimental)
  Interventions: Other: Grape juice R@isol
- grape juice not enriched with polyphenols (Active Comparator)
  Interventions: Other: Commercially-available grape juice

INTERVENTIONS:
Other: Grape juice R@isol
  Arms: Grape juice rich in polyphenols
Other: Commercially-available grape juice
  Arms: grape juice not enriched with polyphenols

SUMMARY:
Many epidemiological and clinical studies have suggested the negative effect of oxidative stress ( = attack of cell components by free radicals) on the cardiovascular risk, notably in patients with metabolic syndrome, insulin resistance, diabetes or obesity and smokers.

Polyphenols, notably those present in red grapes, have a certain antioxidant effect. Dietary supplementation with polyphenols in high-risk patients could diminish the harmful consequences of oxidative stress.

The aim of this study is to show that the daily consumption of grape juice rich in polyphenols " R@isol ", has a positive impact on the oxidation/antioxidation balance in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged from 18 to 50 years
* Men and women
* With national health insurance cover
* With a Body Mass Index between 18.5 and 27.9
* Who have given their written informed consent to take part in the study.

Exclusion Criteria:

* Subjects unable to understand the nature and aims of the study and/or those who have difficulty communicating with the investigator.
* Adults under ward of court.
* Those in custody following a decision of the court or the administration.
* Subjects with a risk of a major change in their diet during the trial.
* Those who drink more than 5 cups of tea or coffee a day.
* Those who consumed more than 25 grammes of alcohol a day, every day of the year preceding the inclusion visit.
* Those who present a history of or current use of psycho-active substances (drugs such as cocain, morphine, heroin...).
* Subjects currently in a period of exclusion relative to another research protocol or for whom the annual cummulation of payments for participation in biomedical research has reached the annual ceiling.
* Presence of any treated chronic disease, and any acute disease within the 4 weeks preceding the inclusion and randomisation visit.
* Persons with diabetes treated with insulin or oral antidiabetics.
* Subjects on lipid-lowering therapy and/or on antioxidants (such as vitamin E, vitamin C, selenium, ß-carotene, Zinc) in the month preceding inclusion.
* Subjects taking multivitamin supplements in the month preceding inclusion.
* Pregnant or breast-feeding women

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2013-10-24 (Actual); Primary Completion 2014-06-17 (Actual); Study Completion 2014-06-17 (Actual)

PRIMARY OUTCOMES:
Measurement of plasma levels of hydroxyoctadecadienoic acid | At inclusion, 15 days and 3 months.

SECONDARY OUTCOMES:
Measurement of endothelial function | At the inclusion and 3 month

CONTACTS AND LOCATIONS:
Locations (1):
- Name CHU Dijon, Dijon, France